CLINICAL TRIAL: NCT03646188
Title: An Open-Label Dose Escalation Trial to Evaluate Dose Limiting Toxicity (DLT), Maximum Tolerated Dose (MTD), Safety, and Tolerability of Microneedle Arrays Containing Doxorubicin (D-MNA) in Participants With Basal Cell Carcinoma (BCC)
Brief Title: Dose Escalation Trial to Evaluate Dose Limiting Toxicity/Maximum Tolerated Dose of Microneedle Arrays Containing Doxorubicin (D-MNA) in Basal Cell Carcinoma (BCC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Application of arrays was inconsistent.
Sponsor: SkinJect, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SKNJCT-001
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Results first posted 2022-08-17 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Intervention Model Description: 3+3 Design
Masking Description: Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo-containing MNA (Placebo Comparator): Placebo
  Interventions: Drug: Placebo-containing MNA
- 25 µg Doxorubicin-containing MNA (Experimental): D-MNA's containing 25 µg of doxorubicin hydrochloride
  Interventions: Drug: 25 µg doxorubicin-containing MNA
- 50 µg Doxorubicin-containing MNA (Experimental): D-MNA's containing 50 µg of doxorubicin hydrochloride
  Interventions: Drug: 50 µg doxorubicin-containing MNA
- 100 µg Doxorubicin-containing MNA (Experimental): D-MNA's containing 100 µg of doxorubicin hydrochloride
  Interventions: Drug: 100 µg doxorubicin-containing MNA
- 200 µg Doxorubicin-containing MNA (Experimental): D-MNA's containing 200 µg of doxorubicin hydrochloride
  Interventions: Drug: 200 µg doxorubicin-containing MNA

INTERVENTIONS:
Drug: Placebo-containing MNA — A 15 x 15 mm array containing 400 tip-loaded, dissolvable microneedles delivering a placebo.
  Other Names: Placebo
  Arms: Placebo-containing MNA
Drug: 25 µg doxorubicin-containing MNA — A 15 x 15 mm array containing 400 tip-loaded, dissolvable microneedles delivering 25 µg of doxorubicin hydrochloride.
  Other Names: 25 µg D-MNA
  Arms: 25 µg Doxorubicin-containing MNA
Drug: 50 µg doxorubicin-containing MNA — A 15 x 15 mm array containing 400 tip-loaded, dissolvable microneedles delivering 50 µg of doxorubicin hydrochloride.
  Other Names: 50 µg D-MNA
  Arms: 50 µg Doxorubicin-containing MNA
Drug: 100 µg doxorubicin-containing MNA — A 15 x 15 mm array containing 400 tip-loaded, dissolvable microneedles delivering 100 µg of doxorubicin hydrochloride.
  Other Names: 100 µg D-MNA
  Arms: 100 µg Doxorubicin-containing MNA
Drug: 200 µg doxorubicin-containing MNA — A 15 x 15 mm array containing 400 tip-loaded, dissolvable microneedles delivering 200 µg of doxorubicin hydrochloride.
  Other Names: 200 µg D-MNA
  Arms: 200 µg Doxorubicin-containing MNA

SUMMARY:
This is a Phase I study in participants with superficial or nodular Basal Cell Carcinoma (BCC), designed to assess dose limiting toxicities and maximum tolerated dose, efficacy, safety, and tolerability of dissolvable, tip-loaded, microneedle arrays containing doxorubicin (D-MNA).

DETAILED DESCRIPTION:
This is a Phase I study in participants with superficial or nodular Basal Cell Carcinoma (BCC), designed to assess dose limiting toxicities and maximum tolerated dose, efficacy, safety, and tolerability of dissolvable, tip-loaded, microneedle arrays containing doxorubicin (D-MNA). Doxorubicin is a cytotoxic anthracycline antibiotic and is currently approved for the treatment of a broad range of cancers, including but not limited to: breast, bladder, gastric, and ovarian cancers; small cell lung cancer; acute lymphoblastic leukemia; and acute myelo blastic leukemia. SkinJect, Inc. has developed a novel delivery system in the form of a tip-loaded dissolvable microneedle array (MNA) which will allow for topical delivery of doxorubicin directly to the lesion at concentrations that are far below standard systemic dosing, thereby reducing the adverse events associated with systemic delivery. The primary objective of this investigation is to establish the highest safe and tolerable dose of single applications of D-MNA, one application per week for three weeks in placebo, 25 µg, 50 µg, 100 µg, and 200 µg dose groups in participants with BCC.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females, 40+ years in general good health as assessed by the investigator.
2. BCC (subtype: superficial or nodular) confirmed histologically by diagnostic shave biopsy at the Screening Visit
3. Primary BCC (i.e., no previous treatment)
4. Lesion size ≥ 4 mm2 or 2 x 2 mm and ≤ 169 mm2 or 13 x 13 mm
5. Participant must have no other "clinically significant" abnormal findings in his/her medical history, physical examination or clinical laboratory test results as assessed by the investigator
6. Negative urine pregnancy at study entry for female of child bearing potential
7. Men and women of child-producing potential must agree to use adequate contraception according to standard instructions by the investigator until the completion of the study
8. Participant must to be willing to adhere to the instructions of the investigator and his or her research team
9. Participant must sign an Informed Consent Form prior to any study specific procedures and entry into the study

Exclusion Criteria:

1. Evidence of clinically significant, unstable medical conditions as assessed by the investigator
2. Excisional biopsy performed on the lesion to be treated in this study
3. Recent therapy(ies) to the BCC treatment area
4. Recurrent BCC (previously treated) at the site presented for treatment
5. BCC lesion to be treated is located in an area where excisional biopsy is undesired or aesthetically unacceptable to the participant
6. Previously demonstrated sensitivity to doxorubicin or carboxymethyl cellulose.
7. Participant with other active malignancies with the exception of non-metastatic prostate cancer and carcinoma in situ of the skin and cervix
8. Concomitant disease requiring systemic immunosuppressive treatment
9. Genetic skin cancer disorder, e.g., basal cell nevus syndrome
10. Participant is pregnant or breastfeeding
11. Treatment with another investigational drug, device, or other intervention within 3 months prior to the Screening Visit
12. Existing condition or treatment within 3 months prior to the Screening Visit that may have impact on clinical outcome for the treatment of BCC or delay in wound healing from the elliptical excision

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Suplick, Study Director — InClinica, Inc.
Locations (1):
- The Center for Clinical and Cosmetic Research, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo-containing MNA | 25 µg Doxorubicin-containing MNA | 50 µg Doxorubicin-containing MNA | 100 µg Doxorubicin-containing MNA | 200 µg Doxorubicin-containing MNA
Started | 3 | 3 | 3 | 3 | 1
Completed | 3 | 3 | 3 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-containing MNA | 25 µg Doxorubicin-containing MNA | 50 µg Doxorubicin-containing MNA | 100 µg Doxorubicin-containing MNA | 200 µg Doxorubicin-containing MNA | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 1 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 0 | 0 | 5
  >=65 years | 2 | 1 | 1 | 3 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.67 (31.72) | 61.33 (8.505) | 63.33 (12.34) | 79 (6.08) | 67 (NA) — There was only 1 subject in this dose cohort. | 67.35 (14.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 1 | 0 | 4
  Male | 3 | 2 | 1 | 2 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 2 | 3 | 1 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 3 | 1 | 13
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities as Assessed by Local Skin Response (LSR) Grading Scale
Description: Dose Limiting Toxicity (DLT) in Trial Subjects Assessed by Local Skin Response Grading Scale, 0-4, 4 being the worst dermal response
Time Frame: 4 weeks
Population: All evaluable subjects
Measure: Number; unit: participants
Arm/Group | Placebo-containing MNA | 25 µg Doxorubicin-containing MNA | 50 µg Doxorubicin-containing MNA | 100 µg Doxorubicin-containing MNA | 200 µg Doxorubicin-containing MNA
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
participants
  Participants | 3 | 3 | 3 | 3 | 1
  Participants with DLTs | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Complete Response (CR) of Eradicated Basal Cell Carcinoma as Measured by Histological Analysis
Description: Complete Response (CR), defined as histological confirmation by central reading of basal cell carcinoma excision in all study participants
Time Frame: 4 weeks
Population: All evaluable subjects
Measure: Number; unit: Participants
Arm/Group | Placebo-containing MNA | 25 µg Doxorubicin-containing MNA | 50 µg Doxorubicin-containing MNA | 100 µg Doxorubicin-containing MNA | 200 µg Doxorubicin-containing MNA
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
Participants | 1 | 2 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: 50 days
Description: Adverse events were recorded throughout the study and at early discontinuation. AEs and medical conditions were coded using the Medical Dictionary for Regulatory Activities (MedDRA) (Version 22.0). Treatment-emergent adverse events (TEAEs) were defined as any event not present prior to the initiation of treatment or any event already present that worsened in either intensity or frequency following exposure to treatment.
Arm/Group | Placebo-containing MNA | 25 µg Doxorubicin-containing MNA | 50 µg Doxorubicin-containing MNA | 100 µg Doxorubicin-containing MNA | 200 µg Doxorubicin-containing MNA
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 0/3 | 0/3 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-containing MNA (N=3) | 25 µg Doxorubicin-containing MNA (N=3) | 50 µg Doxorubicin-containing MNA (N=3) | 100 µg Doxorubicin-containing MNA (N=3) | 200 µg Doxorubicin-containing MNA (N=1)
Application site pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Pain at microneedle array application site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT03646188/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT03646188/SAP_001.pdf